CLINICAL TRIAL: NCT01364480
Title: Microelectrode Brain-Machine Interface for Individuals With Tetraplegia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Boninger (Other)
Responsible Party: Sponsor-Investigator, Michael Boninger, Vice Chair of Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY19030235
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-11

CONDITIONS: Tetraplegia; Spinal Cord Injury
Keywords: Tetraplegia; Spinal cord injury; Brainstem or spinal stroke; Neuroprosthetic; Brain-machine interface; Brain-computer interface; Neural activity
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brain-Machine Interface Users (Experimental): All participants enrolled in the study will undergo Implantation of NeuroPort Arrays in the motor cortex. There is no control group.
  Interventions: Device: Implantation of NeuroPort Arrays in the motor cortex

INTERVENTIONS:
Device: Implantation of NeuroPort Arrays in the motor cortex — Two Blackrock Microsystems NeuroPort Arrays will be implanted in the motor cortex of study participants.
  Other Names: neuroprosthetic; brain-machine interface; brain-computer interface

SUMMARY:
The purpose of this research study is to demonstrate the safety and efficacy of using two NeuroPort Arrays (electrodes) for long-term recording of brain activity.

DETAILED DESCRIPTION:
Individuals with tetraplegia (paralysis caused by illness or injury that results in partial or total loss of use of the arms and legs) have intact brain function but are unable to move due to injury or disease affecting the spinal cord, nerves or muscles. Brain-machine interface (BMI) technology is based on the finding that with intact brain function, neural signals are generated even though they are not sent to the arms, hands and legs. By implanting electrodes in the brain, individuals can be trained to send neural signals which are interpreted by a computer and translated to movement which can then be used to control a variety of devices or computer displays.

ELIGIBILITY:
Inclusion Criteria:

* Limited or no ability to use both hands due to cervical spinal cord injury or brainstem or spinal stroke
* At least 1 year post-injury
* Live within 1 hour of the University of Pittsburgh and be willing to travel to the University of Pittsburgh once per week for BMI training
* Additional inclusion criteria must also be reviewed

Exclusion Criteria:

* Certain implanted devices
* Presence of other serious disease or disorder that could affect ability to participate in this study
* Individuals who are immunosuppressed or who have conditions that typically result in immunocompromise
* Additional exclusion criteria must also be reviewed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2022-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Boninger, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share de-identified data with collaborators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Minimum of seven years after final reporting or publication
Access Criteria: Researchers interested in this topic at the University of Pittsburgh, the University of Chicago, and other centers

REFERENCES:
- [Derived] Sponheim C, Papadourakis V, Collinger JL, Downey J, Weiss J, Pentousi L, Elliott K, Hatsopoulos NG. Longevity and reliability of chronic unit recordings using the Utah, intracortical multi-electrode arrays. J Neural Eng. 2021 Dec 28;18(6):10.1088/1741-2552/ac3eaf. doi: 10.1088/1741-2552/ac3eaf. PMID 34847547
- [Derived] Downey JE, Quick KM, Schwed N, Weiss JM, Wittenberg GF, Boninger ML, Collinger JL. The Motor Cortex Has Independent Representations for Ipsilateral and Contralateral Arm Movements But Correlated Representations for Grasping. Cereb Cortex. 2020 Sep 3;30(10):5400-5409. doi: 10.1093/cercor/bhaa120. PMID 32494819
- [Derived] Downey JE, Schwed N, Chase SM, Schwartz AB, Collinger JL. Intracortical recording stability in human brain-computer interface users. J Neural Eng. 2018 Aug;15(4):046016. doi: 10.1088/1741-2552/aab7a0. Epub 2018 Mar 19. PMID 29553484
- [Derived] Downey JE, Brane L, Gaunt RA, Tyler-Kabara EC, Boninger ML, Collinger JL. Motor cortical activity changes during neuroprosthetic-controlled object interaction. Sci Rep. 2017 Dec 5;7(1):16947. doi: 10.1038/s41598-017-17222-3. PMID 29209023
- [Derived] Downey JE, Weiss JM, Muelling K, Venkatraman A, Valois JS, Hebert M, Bagnell JA, Schwartz AB, Collinger JL. Blending of brain-machine interface and vision-guided autonomous robotics improves neuroprosthetic arm performance during grasping. J Neuroeng Rehabil. 2016 Mar 18;13:28. doi: 10.1186/s12984-016-0134-9. PMID 26987662
- [Derived] Wodlinger B, Downey JE, Tyler-Kabara EC, Schwartz AB, Boninger ML, Collinger JL. Ten-dimensional anthropomorphic arm control in a human brain-machine interface: difficulties, solutions, and limitations. J Neural Eng. 2015 Feb;12(1):016011. doi: 10.1088/1741-2560/12/1/016011. Epub 2014 Dec 16. PMID 25514320
- [Derived] Collinger JL, Wodlinger B, Downey JE, Wang W, Tyler-Kabara EC, Weber DJ, McMorland AJ, Velliste M, Boninger ML, Schwartz AB. High-performance neuroprosthetic control by an individual with tetraplegia. Lancet. 2013 Feb 16;381(9866):557-64. doi: 10.1016/S0140-6736(12)61816-9. Epub 2012 Dec 17. PMID 23253623

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brain-Machine Interface Users
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brain-Machine Interface Users
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Implant
Description: Number of participants who were implanted for at least one year without having to explant the device for safety reasons.
Time Frame: One year following array implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Brain-Machine Interface Users
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: 7 Degree-of-freedom Movement by Neural Control
Description: A modified Action Research Arm Test (ARAT) assessment for upper extremity performance was conducted to evaluate neural control of movement of a robotic prosthetic arm with 7 independent degrees of freedom controlled simultaneously. The degrees of freedom included: 3D translation of arm, 3D orientation of wrist, and 1D open/closing of hand. The participant used a brain-controlled robotic hand to do 9 tasks (out of 19). Each test item was timed and scored as 0 (no movement), 1 (task partly done), 2 (task done, but not correctly), or 3 (task done correctly). Movements that required more than 5 s to complete were scored as 2. The participant attempted each assessment three times and the best score was included. The total possible score ranged from 0 to 27 (i.e., max possible score of 3 each for 9 total tasks). A higher score indicates a better outcome.
Time Frame: One year following array implantation
Measure: Number; unit: score on a scale
Arm/Group | Brain-Machine Interface Users
Number analyzed (Participants) | 1
score on a scale | 16

3. Secondary Outcome: 10 Degree-of-freedom Movement by Neural Control
Description: A modified ARAT was conducted to assess neural control of movement of a robotic prosthetic arm with 10 independent degrees of freedom, controlled simultaneously. Degrees of freedom included: 3D translation of arm, 3D orientation of wrist, and 4 degrees dictating hand shape, including pinch (flexion of thumb, index and middle fingers), scoop (flexion of ring and pinky fingers), finger abduction (of index, ring and little fingers), and thumb opposition. The participant used a brain-controlled robotic hand to do 9 tasks (out of 19). Test items were timed and scored as 0 (no movement), 1 (task partly done), 2 (task done, but not correctly), or 3 (task done correctly). Movements that required more than 5 s to complete were scored as 2. The participant attempted each assessment three times and the best score was included. The total possible score ranged from 0 to 27 (i.e., max possible score of 3 each for 9 total tasks). A higher score indicates a better outcome.
Time Frame: One year following array implantation
Measure: Number; unit: score on a scale
Arm/Group | Brain-Machine Interface Users
Number analyzed (Participants) | 1
score on a scale | 15.6

ADVERSE EVENTS:
Time Frame: through study completion, 2 years, 8.5 months duration of implant
Groups:
- Brain-Machine Interface Users: All eligible participants enrolled in the study will undergo Implantation of NeuroPort Arrays in the motor cortex. There is no control group.
  Two Blackrock Microsystems NeuroPort Arrays will be implanted in the motor cortex of study participants.
Arm/Group | Brain-Machine Interface Users
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brain-Machine Interface Users (N=1)
Skin retraction at pedestal site (Skin and subcutaneous tissue disorders) | 1 (1) — Around percutaneous pedestal sites on the scalp, skin started pulling away from the pedestals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT01364480/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT01364480/ICF_001.pdf